CLINICAL TRIAL: NCT01991028
Title: An Open Label, Randomised, Two-way Crossover Scintigraphic Study to Investigate Lung Deposition of Radiolabelled OligoG Delivered as a Dry Powder and as a Nebulised Solution in Cystic Fibrosis Patients
Brief Title: A Study to Investigate Lung Deposition of Radiolabelled OligoG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BDD Pharma Ltd (Industry)
Collaborators: AlgiPharma AS (Industry)
Responsible Party: Principal Investigator, Howard Stevens, Principal Investigator, BDD Pharma Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BC-180-12
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiolabelled OligoG CF-5/20 DPI (Experimental): Single dose OligoG CF-5/20 Dry Powder for Inhalation by 3 capsules of 32mg OligoG via Miat Monodose Inhaler, radiolabelled ca10MBq 99mTc.
  Interventions: Drug: Radiolabelled OligoG CF-5/20 DPI
- Radiolabelled OligoG CF-5/20 6% Solution (Active Comparator): Single dose of 1.5mL (90mg) aerosolised OligoG CF-5/20 6% solution via Sidestream Plus nebuliser, radiolabelled ca10MBq 99mTc.
  Interventions: Drug: Radiolabelled OligoG CF-5/20 6% Solution

INTERVENTIONS:
Drug: Radiolabelled OligoG CF-5/20 DPI — Inhalation with dry powder by Mia Monodose Inhaler
  Other Names: Radiolabelled OligoG CF-5/20 Dry Powder for Inhalation
  Arms: Radiolabelled OligoG CF-5/20 DPI
Drug: Radiolabelled OligoG CF-5/20 6% Solution — Inhalation with aerosolised solution by nebuliser
  Other Names: Radiolabelled OligoG CF-5/20 Solution
  Arms: Radiolabelled OligoG CF-5/20 6% Solution

SUMMARY:
OligoG is a new potential treatment which is being developed by AlgiPharma AS (a Norwegian-based company) with an aim to help people with cystic fibrosis in the future.

OligoG, derived from marine algae, is expected to act locally in the lungs once inhaled to reduce mucus thickness and improve mucus clearance. It could also have the benefit of reducing the incidence of infections.

Nebulised doses of up to 540 mg/day have been administered to healthy volunteers for three consecutive days and to cystic fibrosis patients for 28 consecutive days. Both groups tolerated the medication well, with no treatment related issues reported. The dose administered in this study is lower; patients who complete the study will receive, in total, 186 mg of OligoG in two divided doses.

A new dry powder formulation of OligoG has been developed so that patients can use an inhaler, rather than a nebuliser. Administration from an inhaler compared to a nebuliser is much quicker and more practical for the patient.

In this study, we will use gamma scintigraphy to see where in the lungs the dry powder and nebulised solution go after being inhaled by cystic fibrosis patients. Gamma scintigraphy is a well-established medical imaging technique. A small amount of radioactive material will be added to both the dry powder and nebulised solution. The radiation emitted will then be detected by taking images using a device known as a gamma camera. The procedure is relatively easy and non-invasive.

The purpose of this study is to help answer the following research questions:

* How do the OligoG dry powder and nebulised solution distribute in the lungs of patients with cystic fibrosis?
* How much of the formulation gets to the deep lung?
* How much of the formulation remains in the devices used for administration?

DETAILED DESCRIPTION:
The primary efficacy (deposition) variable will be the % dose deposited in the lungs.

The following secondary efficacy (deposition) variables will be determined (where appropriate): Percentage dose deposited in the oropharyngeal, oesophageal and gastric regions Percentage dose remaining in the Miat Monodose inhaler Percentage dose remaining in the nebuliser mouthpiece Percentage dose remaining in the nebuliser reservoir Percentage dose deposited on the exhalation filter (if appropriate) Percentage dose contained in mouth washing(s) Penetration index based on the ratio of counts in the central:peripheral lung regions (C/P index)

ELIGIBILITY:
Inclusion Criteria:

Aged at least 18 years at screening. Understands and is willing, able and likely to comply with all study procedures and restrictions.

Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any trial-related activities.

Male or female with a confirmed diagnosis of cystic fibrosis defined by:

i.Clinical features consistent with the diagnosis of cystic fibrosis (Rosenstein et al., 1998); AND ii.Sweat chloride ≥ 60 mmol/L by pilocarpine iontophoresis; OR iii.Genotypic confirmation of 2 CF-causing mutations

Positive microbiological finding of Pseudomonas aeruginosa (mucoid or nonmucoid) in expectorated sputum (and/or swab) documented within the last 24 months prior to screening. Negative finding is acceptable provided the proportion of patients enrolled with positive findings is at least 80%.

At screening, FEV1 must be between 35 and 80% of the predicted normal value following adjustment for age, gender and height according to the Knudson equation (Knudson et al., 1983)

Clinically stable in the opinion of the referring physician at CF unit.

Female subjects of child-bearing potential and male subjects participating in the study who are sexually active must use acceptable contraception. For the purpose of this study, acceptable contraception is defined as:

i.Oral, injected or implanted hormonal methods or contraception; OR ii.Placement of an intrauterine device (IUD) or intrauterine system (IUS); OR iii.Barrier methods of contraception: condom or occlusive cap with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

On-going acute illness. Patients must not have needed an outpatient visit, hospitalisation or required any change in therapy for other pulmonary disease between screening and AV1.

History of, or planned organ transplantation.

Requirement for continuous (24 hour/day) oxygen supplementation.

Concomitant administration of inhaled mannitol or hypertonic saline within 48 hours of Period 1, Day 1.

Clinically significant abnormal findings on haematology or clinical chemistry. In addition, any value ≥ 3 x the upper limit of normal will exclude the patient from participating in the study.

Unable to perform pulmonary function tests according to ATS criteria.

Pregnant or breast-feeding women.

Participated in any interventional clinical trial within the 28 days prior to AV1.

Documented or suspected, clinically significant, alcohol or drug abuse.

Known allergies or intolerances to alginates.

Any active malignant disease (with the exception of basal cell carcinoma; BCC).

Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol.

Haemoptysis more than 60 mL at any time within 30 days before study drug administration.

Participation in this study will exceed the limits of total radiation exposure allowed in any 12 month period (5 mSv), or will exceed 10 mSv over any three year period.

Males who intend to father a child in 3 months following study or are unwilling to abstain from sexual intercourse with pregnant or lactating women. Females who are intending to become pregnant in 3 months following study.

Any non-removable metal objects such as metal plates, screws etc in their head, neck, chest or abdominal area.

As a result of a physical examination or screening investigations, the physician responsible considers the patient unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To qualitatively determine the deposition of radiolabelled OligoG in the lung. | 1 day (Scintigraphic imaging will be performed at one time point only; immediately after dosing)

SECONDARY OUTCOMES:
To determine the radiolabel distribution pattern of the two formulations in the diseased lung, including calculating the ratio of radiolabel in the central airways compared to the peripheral region (C/P index) | 1 day (Scintigraphic imaging will be performed at one time point only; immediately after dosing)
To characterise the extrapulmonary deposition (i.e. oropharyngeal and stomach) of radiolabel including retention in the nebuliser or dry powder inhaler reservoir and deposition on the exhalation filter (if appropriate) | 1 day (Scintigraphic imaging will be performed at one time point only; immediately after dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Howard NE Stevens, PhD, Principal Investigator — BDD Pharma Ltd
Locations (1):
- Bio-Images Research Ltd, Glasgow, United Kingdom